CLINICAL TRIAL: NCT03420118
Title: Molecular and Immunological Characterization of Gynecological Malignancies
Brief Title: Study of Biomarkers in Gynecological Cancers
Acronym: VENUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VENUS; 17-5411 (Other: UHN REB)
Record Dates: First submitted 2017-11-16; First posted 2018-02-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor tissue and blood samples collection (Experimental)
  Interventions: Procedure: Tumour tissue collection; Procedure: Blood draws

INTERVENTIONS:
Procedure: Tumour tissue collection — Depending on the status of disease when participants join the study, a sample of tumour tissue may be collected from:
  * A previous surgery for the disease,
  * A biopsy for diagnosing the disease,
  * Other surgical procedures done for clinical management or possible cancer related complications (e.g., bowel obstruction).
  In addition:
  * Patients undergoing pre-screening prior to diagnosis will have tumour sample collected at the time of surgery.
  * At anytime participants require a biopsy as a part of their cancer care, a sample of that tumour tissue will be collected.
  * New biopsies will be done to collect fresh tumour tissue each time participants' disease worsens.
Procedure: Blood draws — Blood samples will be collected at the following different times points:
  * All patient undergoing pre-screening for histological diagnosis will have blood samples collected.
  * Before starting a new line of treatment for the disease,
  * One week after starting a new line of treatment for the disease,
  * During treatment, at each radiological assessment (imaging scan) that will be done to check the status of the disease,
  * At the time the disease worsens or relapses (comes back)
  * During observation/follow-up, at the time of any radiological assessments that will be done to check the status of the disease

SUMMARY:
In recent years, there has been a significant improvement in understanding the biology of cancer and this information has been used to improve cancer care and patient outcome.

Research has shown that changes in some genes and/or proteins may be important indicators for certain cancers and response to treatments. Genes are molecules made up of ribonucleic acid (RNA) and deoxyribonucleic acid (DNA). DNA contain instructions for the development and functioning of the cells in the body and are passed down from parent to child. RNA is involved with producing proteins in the body. Further research is needed to better understand the changes found in cancer cells and how to target them to stop or reduce cancer growth.

A drug that may be able to block certain specific cancer cell changes is called "targeted therapy". Different people with the same type of cancer receiving the same drug could have different responses to it. For example, one person may experience a reduction of their tumor while another person's cancer may worsen. The reason for this is still not well understood and could lie in gene changes.

Understanding these changes may allow researchers to predict how treatments may work in guiding decisions around choice of drugs.

The purpose of the study is to learn more about gene changes or protein expression (levels) of tumors to better understand the behavior of gynecological diseases and, if possible, better address participants' cancer care now or in the future.

ELIGIBILITY:
Pre-Screening Eligibility:

Inclusion Criteria:

* Patients with probable diagnoses of gynecological malignancy (ovarian, tubal, primary peritoneal, uterine, cervical, vulvar and rare gynecological cancers) and confirmed to be undergoing upfront debulking surgery/radiation
* Patient must be ≥16 years of age at the time of consent.
* Ability to understand and provide written informed consent.
* ECOG Performance Status ≤ 2.
* Patient must consent to provide tissue sample from surgery and blood samples
* Life expectancy ≥3 months.

Exclusion Criteria:

* Patients must be treatment naïve (no previous treatment of Neoadjuvant chemotherapy nor radiation for newly diagnosed disease)

Eligibility for Patients with Gynecological Diagnosis

Inclusion Criteria:

* Patients with histological confirmation of gynecological malignancy (except ovarian cancer with high grade serous histology, tubal, primary peritoneal, uterine, cervical, vulvar and vaginal cancer and rare gynecological cancers).
* Patient must be ≥16 years of age at the time of consent.
* Ability to understand and provide written informed consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Patient must consent to providing archival tissue and/or to undergo tumour biopsy and/or to provide blood or fluid collection samples. Patients will also be asked to provide a blood sample for germline mutation analysis.
* Life expectancy ≥3 months.
* No limits of previous lines of treatment.

Exclusion Criteria:

* Any contraindication to tumour biopsy or blood collection
* Patient with diagnosis of High grade serous Ovarian Cancer are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2027-12-21 (Estimated)

PRIMARY OUTCOMES:
Genomic and immune signatures in terms of progression free survival | 5 years
Genomic and immune signatures in terms of overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No